CLINICAL TRIAL: NCT00542022
Title: A Placebo-Controlled, Parallel-Group, Double-Blind, 12-Week Study to Assess the Clinical Efficacy, Safety, and Tolerability of MK0812 in Rheumatoid Arthritis Patients
Brief Title: Efficacy, Tolerability and Safety Study in Rheumatoid Arthritis (0812-008)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0812-008; MK0812-008; 2007_631
Record Dates: First submitted 2007-10-05; First posted 2007-10-10 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-10

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Duration of Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0812 / Duration of Treatment: 12 Weeks
Drug: Comparator: placebo (unspecified) / Duration of Treatment: 12 Weeks

SUMMARY:
To demonstrate the clinical effectiveness of MK0812 in the treatment of Arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Patient has had diagnosis of RA made at least 6 months prior to study start and was greater than 16 years of age when diagnosed
* Patient has active RA with a minimum level of disease activity including at least 10 swollen joints and 10 tender or painful joints
* Excepting rheumatoid arthritis, patient is judged to be in otherwise general good health based on medical history, physical examination, and routine laboratory tests

Exclusion Criteria:

* Patient is mentally or legally incapacitated, has significant emotional problems at the time of the study, or has a history of psychosis
* Patient has a history of any clinically significant disease of the cardiovascular, hepatic, neurological, renal, genitourinary, or hematologic systems or uncontrolled blood pressure
* Female patient is pregnant or breast-feeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2004-06; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
MK0812 once daily for 12 weeks will demonstrate clinical effectiveness superior to placebo for treatment of Arthritis, as assessed by changes from baseline in the patient's swollen joint count | 12 weeks

SECONDARY OUTCOMES:
MK0812 once daily for 12 weeks will be safe and well tolerated in Arthritis patients | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC